CLINICAL TRIAL: NCT00978354
Title: A Phase II Randomized Blinded Controlled Trial of the Effect of furoSemide in Critically Ill Patients With eARly Acute Kidney Injury (The SPARK Study)
Brief Title: Furosemide in Early Acute Kidney Injury
Acronym: SPARK
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Feasibility of target enrollment within the context of available funding resources.
Sponsor: University of Alberta (Other)
Collaborators: Austin Hospital, Melbourne Australia (Other); Princess Alexandra Hospital, Brisbane, Australia (Other)
Responsible Party: Principal Investigator, Sean M Bagshaw, Associate Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHFMR-0920
Record Dates: First submitted 2009-09-14; First posted 2009-09-16 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Acute Renal Failure
Keywords: acute kidney injury; acute renal failure; loop diuretic; critical illness; sepsis; renal replacement therapy; dialysis; renal recovery; survival
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness; Sepsis | interventions — Furosemide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Furosemide (Active Comparator): Furosemide intravenous continuous infusion
  Interventions: Drug: Furosemide
- Normal Saline (Placebo Comparator): Normal saline titrated continuous intravenous infusion
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Furosemide — Continuous intravenous infusion of furosemide titrated to urine output
  Other Names: Lasix
  Arms: Furosemide
Drug: Normal Saline — Continuous intravenous infusion 0.9% normal saline placebo control
  Other Names: 0.9% saline
  Arms: Normal Saline

SUMMARY:
Acute renal failure, now referred to as acute kidney injury, is common in intensive care unit patients, contributes to high morbidity and mortality, and has no proven interventions with benefit once established. In addition to supportive care, these patients frequently receive diuretic therapy, most commonly furosemide.

Prior trials showed no impact of furosemide on clinical outcomes and perhaps harm, however, these trials suffered from numerous limitations and lack applicability to modern intensive care unit patients. As a result, there appears a disconnect between clinical practice and available evidence. Survey data supports the view of clinical equipoise for use of furosemide in intensive care unit patients with early acute kidney injury. Moreover, these data also confirm there is an urgent need for higher quality and more definitive evidence from randomized trial on furosemide use in early acute kidney injury.

Accordingly, the investigators propose to conduct a pilot phase II randomized, blinded, placebo-controlled trial comparing furosemide to placebo in ICU patients with early acute kidney injury.

The specific aims of this study are:

1. To compare the efficacy and safety of a continuous infusion of furosemide versus placebo titrated to the physiology parameter of urine output in early acute kidney injury on the primary outcome of progression in severity of kidney injury in intensive care unit patients with early AKI and stratified by the presence of sepsis.
2. To evaluate selected secondary endpoints on the impact of furosemide versus placebo, specifically: fluid balance goals; electrolyte and acid-base balance; the need for renal replacement therapy (i.e. dialysis); total duration of acute kidney injury; the rate of renal recovery; and mortality.
3. To compare the impact of furosemide versus placebo on the trajectory of serum and urinary biomarkers (neutrophil gelatinase-associated lipocalin [NGAL], interleukin-18 [IL-18]) and evaluate whether these biomarkers perform superior to conventional measures (creatinine, urea) for monitoring the progression of kidney injury and the prediction of outcome.

This trial represents part of a larger initiative aimed towards expanding our understanding of the treatment of acute kidney injury in intensive care unit patients and evaluating interventions that may potentially reduce kidney injury and improve clinical outcomes.

DETAILED DESCRIPTION:
Study Design, Setting and Patient Population

This is a phase II multi-centre, randomized, blinded, placebo-controlled trial of ICU patients with early AKI with randomization stratified by sepsis. All critically ill patients admitted to the participating ICUs will be screened for eligibility.

Operational Definitions

1. Acute kidney injury (AKI) - The operational definition for early AKI will be defined and classified according to the RIFLE criteria (and modified AKIN). The presence of early AKI will be defined by the RIFLE class - RISK: an abrupt (within 48hr) reduction in kidney function characterized by an relative increase in serum creatinine of >50% (1.5 fold) or >26.5 mcmol/L from baseline or a reduction in urine output of ≤0.5 mL/kg/hr for >6 hours.

Trial Protocol

Description of Study Flow

Patients will be identified in the ICU by daily surveillance of admitted patients by the PI and/or research coordinator or when identified by the treating ICU physician. Each patient's eligibility will be verified by use of a one-page checklist that summarizes the inclusion and exclusion criteria. This checklist will be included in the standardized case-report form (CRF).

Study Intervention

Following obtainment of consent, patients will be commenced on a continuous infusion of either the intervention (furosemide) or identical placebo (0.9% NaCl). The study protocol for administration of furosemide by continuous infusion is adapted from the phase I study by Ostermann et al. The study infusion bag will contain 2000mg of furosemide in 500mL of 0.9%NaCl for a final concentration of 4mg/mL. The continuous infusion will be titrated to achieve a target urine output in the range of 1.0-2.0 mL/kg/hr. Each patient will be administered a loading dose of 0.4 mg/kg as a separate infusion bag followed by a continuous infusion commenced at a dose of 0.0125 ml/kg/hr. The maximum infusion rate will be 0.125ml/kg/hr. The urine output will be assessed hourly. If the target urine output has been achieved, then the current infusion rate will be continued. If the target urine output has not been achieved, the dose will be increased to the next infusion rate in the algorithm. If the urine output is too brisk (>2mL/kg/hr), the dose will be maintained unless any of the following criteria are fulfilled: decrease in mean arterial pressure <65 AND/OR addition of or an increase in vasoactive requirements of ≥20% to achieve goal mean arterial pressure OR central venous pressure <8 cmH2O OR central venous oxygen saturation <60% OR a cardiac index <2.0L/min/1.73m2 (if measured). If any of these criteria are achieved, the dose will be decreased to the next lower infusion rate in the algorithm. If any of the aforementioned criteria have been fulfilled AND urine output remains >2mL/kg/hr for 2 consecutive hours despite the lowest infusion rate, the treatment will be discontinued for 1 hour then resumed at the lowest infusion rate. The fulfillment of these criteria will be brought to the attention of the consultant ICU physician for review. At any time during the trial, if the responsible ICU physician believes that diuretics are urgently indicated (pulmonary edema), diuretics can be administered and this event will be documented.

All other aspects of patient management within the parameters outlined (methods of fluid resuscitation, choice of fluids, vasoactive therapy, choice of vasoactive therapy, adjuvant therapies such as hrAPC, intensive insulin therapy, will be at the discretion of the consultant ICU physician.

The study drug infusion will be continued until any one of the following events occur:

1. the patient is initiated on RRT;
2. the patient dies;
3. the patient is discharged from the ICU;
4. the patient recovers kidney function; or
5. the patient develops a recognized adverse reaction potentially related to the study infusion.

Methods of Randomization

The randomization sequence will be created at a single central location at the University of Alberta Hospital (EPICORE Centre). The sequence will be stratified by the presence of a diagnosis of sepsis.

Data Collection

Detailed clinical, physiologic, laboratory and outcome data will be collected. Data will be collected each day on whether the primary endpoint (progression of AKI) has occurred, for evidence of any secondary endpoints and criteria for trial discontinuation. Plasma and urine will be collected for biomarkers studies. Any study protocol violations will be recorded. The adjudication of protocol violations will be determined by a study investigator blinded to the treatment allocation.

Proposed Follow-up

The investigators plan to follow all patients to determine the duration of AKI, continued need for RRT, renal recovery and mortality until death or discharge from hospital and at 30, 60 and 90-days after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Informed and written consent by patient or surrogate
* Peripheral or central intravenous catheter
* The presence of early AKI
* 2 or more criteria for the systemic inflammatory response syndrome (SIRS) within 24 hours
* Achieved immediate resuscitation goals

Exclusion Criteria:

* Confirmed or suspected pregnancy
* Age <18 years
* Stage 4 or greater chronic kidney disease or kidney transplantation
* Acute pulmonary edema requiring urgent use of furosemide or RRT
* Patient is moribund with expected death within 24 hours
* Known or suspected drug allergy to furosemide
* Enrolled in concomitant randomized trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-09; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Worsening AKI | 7 days

SECONDARY OUTCOMES:
Fluid balance | 7 days
Renal replacement therapy (RRT) | 7 days
Renal Recovery | 90-days
Survival | 90-days

CONTACTS AND LOCATIONS:
Overall Officials: Sean M Bagshaw, MD MSc, Principal Investigator — University of Alberta
Locations (4):
- Australia (2):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Austin Hospital, Melbourne, Victoria
- Canada (2):
  - General Systems Intensive Care Unit, University of Alberta, Edmonton, Alberta
  - University of Laval, Québec, Quebec

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152
- [Derived] Bagshaw SM, Gibney RTN, Kruger P, Hassan I, McAlister FA, Bellomo R. The effect of low-dose furosemide in critically ill patients with early acute kidney injury: A pilot randomized blinded controlled trial (the SPARK study). J Crit Care. 2017 Dec;42:138-146. doi: 10.1016/j.jcrc.2017.07.030. Epub 2017 Jul 12. PMID 28732314
- [Derived] Bagshaw SM, Gibney RT, McAlister FA, Bellomo R. The SPARK Study: a phase II randomized blinded controlled trial of the effect of furosemide in critically ill patients with early acute kidney injury. Trials. 2010 May 11;11:50. doi: 10.1186/1745-6215-11-50. PMID 20459801